CLINICAL TRIAL: NCT00354016
Title: A Phase III, Multicenter, Uncontrolled, Open-Label Study to Demonstrate Safety and Immunogenicity of a Commercially Available Preservative Free Inactivated Split Influenza Vaccine, Using the Strain Composition 2006/2007 When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Preservative Free Inactivated Split Influenza Vaccine, Using the Strain Composition 2006/2007 in Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V44P10S; EudraCT number 2006-000438-11
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Influenza
Keywords: influenza; vaccine
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: preservative free inactivated split influenza vaccine using the strain composition 2006/2007

SUMMARY:
Due to antigenic changes of influenza viruses, the virus strains used in influenza vaccines are adjusted every year according to WHO (World Health Organization) and CHMP (Committee for Medicinal Products for Human Use) recommendations. Immunogenicity and tolerability of the newly composed vaccines are subject for evaluation in a yearly clinical trial in non-elderly and elderly subjects (CPMP/BWP/214/96).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged >18 years

Exclusion Criteria:

* serious chronic diseases or significant acute infections requiring systemic antibiotic treatment
* history of any anaphylaxis, serious vaccine reactions
* hypersensitivity against vaccine components
* history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* known or suspected impairment/alteration of immune function
* more than one injection of influenza vaccine received or laboratory confirmed influenza disease
* within last 6 months: influenza vaccination received

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2006-07

PRIMARY OUTCOMES:
antibody titers to each influenza strain measured by hemagglutination inhibition (HI) test on Day 0 and on Day 21

SECONDARY OUTCOMES:
safety of a single IM dose of the split influenza vaccine using solicited local and systemic reactions and adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Chair — Novartis Vaccines & Diagnostics
Locations (2):
- Germany (2):
  - Werksarztzentrum Herborn, Westerwaldstr 36,, Herborn
  - Betriebsarztlicher Dienst, Universitat Marburg, Robert-Koch-Str, 5,, Marburg